CLINICAL TRIAL: NCT03155347
Title: A Randomized, Multi-Center, Double Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Subcutaneous (SC) Tocilizumab (TCZ) in Combination With Methotrexate (MTX) and as Monotherapy Versus MTX in Patients With Moderate to Severe Rheumatoid Arthritis With Inadequate Response to Current DMARD Therapy
Brief Title: An Efficacy and Safety Study of Subcutaneous Tocilizumab in Combination With Methotrexate (MTX) and as Monotherapy Versus MTX in Participants With Moderate to Severe Rheumatoid Arthritis With Inadequate Response to Current Disease-Modifying Antirheumatic Drug (DMARD) Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YA29359
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tocilizumab + MTX (Experimental): Participants will receive tocilizumab SC injections Q2W along with MTX orally every week (QW) for 24-week double-blind treatment phase. Participants who complete the 24-week double-blind treatment phase may continue treatment until Week 48 in the extension phase, irrespective if they achieve or do not achieve DAS28 low activity (DAS28-ESR <= 3.2).
  Interventions: Drug: Tocilizumab; Drug: MTX
- Tocilizumab + Placebo Matched to MTX (Experimental): Participants will receive tocilizumab SC Q2W along with placebo matched to MTX for 24-week double-blind treatment phase. Participants who complete the 24-week double-blind treatment phase may continue treatment until Week 48 in the extension phase. In the extension phase up to Week 48, participants who achieve DAS28 low activity (DAS28-ESR <= 3.2) will remain on the same treatment they received in double-blind phase. Participants who do not achieve DAS28-ESR <= 3.2 will receive treatment with tocilizumab 162 mg SC Q2W + MTX from Week 26 to Week 48.
  Interventions: Drug: Tocilizumab; Drug: MTX; Drug: Placebo Matched to MTX
- Placebo Matched to Tocilizumab + MTX (Active Comparator): Participants will receive placebo matched to tocilizumab along with MTX orally QW for 24-week double-blind treatment phase. Participants who complete the 24-week double-blind treatment phase may continue treatment until Week 48 in the extension phase. In the extension phase up to Week 48, participants who achieve DAS28 low activity (DAS28-ESR <= 3.2) will remain on the same treatment they received in double-blind phase. Participants who do not achieve DAS28-ESR <= 3.2 will receive treatment with tocilizumab 162 mg SC Q2W + MTX from Week 26 to Week 48.
  Interventions: Drug: Tocilizumab; Drug: MTX; Drug: Placebo Matched to Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive tocilizumab 162 mg given as 0.9 milliliter (mL) of a 180 mg/mL solution in a prefilled syringe, administered by SC injection Q2W.
  Other Names: RO4877533
Drug: MTX — Participants will receive MTX stable doses at 10 to 25 mg orally.
Drug: Placebo Matched to MTX — Placebo matched to MTX.
  Arms: Tocilizumab + Placebo Matched to MTX
Drug: Placebo Matched to Tocilizumab — Placebo matched to tocilizumab.
  Arms: Placebo Matched to Tocilizumab + MTX

SUMMARY:
This is a randomized, double-blind, multi-center, parallel-group study to evaluate the efficacy and safety of subcutaneous (SC) tocilizumab (162 milligrams [mg] every 2 weeks [Q2W]) given as monotherapy and in combination with MTX versus MTX given as monotherapy, in participants with moderate to severe active rheumatoid arthritis (RA) who have inadequate response to current DMARD therapy. The study comprises a 24-week double-blind treatment phase, followed by a 24-week extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participants who are located in mainland China with RA of greater than or equal to (>=) 6 months' duration from onset of the disease, diagnosed according to the revised 1987 ACR criteria and receiving treatment on an outpatient basis
* Participants must have discontinued etanercept (or YiSaiPu) for >= 2 weeks, infliximab, certolizumab, golimumab, abatacept or adalimumab for >= 8 weeks, anakinra for >= 1 week prior to randomization
* Have received oral MTX at a stable dose for at least 12 weeks prior to baseline (MTX dose 10 to 25 mg) and experience of failing at least one non-biologic DMARD including MTX
* All treatment with non-biological DMARDs except MTX should be withdrawn at least 2 weeks prior to baseline (leflunomide for >= 12 weeks or >= 14 days after standard cholestyramine or activated charcoal washout, azathioprine for >= 4 weeks)
* SJC >= 6 (on the basis of 66 joint counts) and TJC >= 8 (on the basis of 68 joint counts) at screening and baseline with at least 3 months of treatment with permitted DMARDs
* Participants must have either high sensitive CRP >= 10 milligrams per liter (mg/L) or ESR >=28 millimeters per hour (mm/hr) at screening
* Oral corticosteroids (<=10 mg/day prednisone or equivalent) and nonsteroidal anti-inflammatory drug (NSAIDs; up to the maximum recommended dose per local standard of care) are permitted if the dose has been stable for at least 4 weeks prior to baseline
* All treatment with Chinese traditional medicine and/or herb medicine for RA treatment should be withdrawn at least 2 weeks prior to baseline
* Females of childbearing potential and males with female partners of childbearing potential may participate only if using a reliable means of contraception as defined by the protocol

Exclusion Criteria:

* Participants with major surgery or planned major surgery, rheumatic autoimmune disease other than RA, and functional class IV (as defined by the ACR Classification of Functional Status in RA)
* Participants with unsuccessful treatment with an anti-tumor necrosis factor (anti-TNF) agent; previous treatment with any cell-depleting therapies including investigational agents and janus kinase (JAK) inhibitors or any other new agents which have DMARD/DMARD-like effect; treatment with intravenous (IV) gamma-globulin, plasmapheresis, or Prosorba column; treatment with alkylating agents
* Intra-articular or parenteral corticosteroids and/or immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of serious uncontrolled concomitant diseases and disease states; evidence of active malignant disease
* Participants with abnormal haematological parameters, abnormal renal and hepatic parameters
* Positive for either hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and/or hepatitis C virus (HCV) antibody

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology (ACR) 20 (ACR20) Response at Week 24 | Week 24

SECONDARY OUTCOMES:
Percentage of Participants With Low Disease Activity at Week 24, Defined as Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR) Score of Less Than or Equal to (<=) 3.2 | Week 24
Percentage of Participants With Remission at Week 24, Defined as DAS28-ESR Score of Less Than (<) 2.6 | Week 24
Change From Baseline in Tender Joint Count (TJC) at Week 24 | Baseline, Week 24
Change From Baseline in Swollen Joint Count (SJC) at Week 24 | Baseline, Week 24
Change From Baseline in C-reactive Protein (CRP) Levels at Week 24 | Baseline, Week 24
Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 24 | Baseline, Week 24
Change From Baseline in the Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS) Score at Week 24 | Baseline, Week 24
Change From Baseline in the Physician's Global Assessment of Disease Activity VAS Score at Week 24 | Baseline, Week 24
Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24 | Baseline, Week 24
Change From Baseline in the Patient's Pain VAS at Week 24 | Baseline, Week 24
Change From Baseline in DAS28-ESR at Week 24 | Baseline, Week 24
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 56 weeks
Percentage of Participants With anti-Tocilizumab Antibody | Baseline, Week 12, Week 24, Week 48, at the time of withdrawal up to approximately 48 weeks
Serum Interleukin-6 (IL-6) Levels | Baseline, predose (Hour 0) on Weeks 2, 4, 8, 12, 16, 24, 48
Serum Soluble Interleukin-6 Receptor (sIL-6R) Levels | Baseline, predose (Hour 0) on Weeks 2, 4, 8, 12, 16, 24, 48
Maximum Observed Plasma Concentration (Cmax) of Tocilizumab | predose (Hour 0) and 6-hours postdose on Day 0, Day 84; predose (Hour 0) on Day 14 and 98; on Day 1, 2, 3, 5, 7, 10, 85, 86, 87, 89, 91, and 94
Minimum Observed Plasma Concentration (Cmin) of Tocilizumab | predose (Hour 0) on Day 0, 14, 84, and 98; on Day 1, 2, 3, 5, 7, 10, 85, 86, 87, 89, 91, and 94
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Tocilizumab | predose (Hour 0) and 6-hours postdose on Day 0, Day 84; predose (Hour 0) on Day 14 and 98; on Day 1, 2, 3, 5, 7, 10, 85, 86, 87, 89, 91, and 94
Plasma Decay Half-Life (t1/2) of Tocilizumab | predose (Hour 0) and 6-hours postdose on Day 0, Day 84; predose (Hour 0) on Day 14 and 98; on Day 1, 2, 3, 5, 7, 10, 85, 86, 87, 89, 91, and 94
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) of Tocilizumab | predose (Hour 0) and 6-hours postdose on Day 0, Day 84; predose (Hour 0) on Day 14 and 98; on Day 1, 2, 3, 5, 7, 10, 85, 86, 87, 89, 91, and 94
Accumulation Ratio for Area Under the Concentration Time Curve (Rac, AUC) of Tocilizumab | predose (Hour 0) and 6-hours postdose on Day 0, Day 84; predose (Hour 0) on Day 14 and 98; on Day 1, 2, 3, 5, 7, 10, 85, 86, 87, 89, 91, and 94
Accumulation Ratio for Maximum Observed Plasma Concentration (Rac, Cmax) of Tocilizumab | predose (Hour 0) and 6-hours postdose on Day 0, Day 84; predose (Hour 0) on Day 14 and 98; on Day 1, 2, 3, 5, 7, 10, 85, 86, 87, 89, 91, and 94
Accumulation Ratio for Minimum Observed Plasma Trough Concentration (Rac, Cmin) of Tocilizumab | predose (Hour 0) on Day 14, 84
Plasma Trough Concentration (Ctrough) of Tocilizumab | predose (Hour 0) on Day 0, 14, 28, 56, 84, 98, 112, 140, 168, and 336
Percentage of Participants With ACR50 Responses at Week 24 | Week 24
Percentage of Participants With ACR70 Responses at Week 24 | Week 24

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Union Hospital, Beijing
  - Affiliated Hospital of Bengbu Medical College, Bengbu
  - the First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong General Hospital, Guangzhou
  - The 1st Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Affiliated Hospital of Inner Mongolia Medical College, Hohhot
  - The First Hospital of Jiaxing, Jiaxing
  - Qilu Hospital of Shandong University, Jinan
  - The First Affilliated Hospital of Kunming Medical College, Kunming
  - Jiangsu Province Hospital, Nanjing
  - Pingxiang People Hospital, Pingxiang
  - Shengjing Hospital of China Medical University, Shenyang
  - The Second Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu T, Wang L, Zhang X, Chen L, Liu Y, Jiang Z, Shuai Z, Zhang M, Wei W, Liu H, Xu J, Zhang Z, Wang G, Wang X, Hu J, Li H, Zhang Z, Wang H, Lu F, Du Y, Xue Z, Zhao Y, Li Z. Tocilizumab Monotherapy or Combined With Methotrexate for Rheumatoid Arthritis: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2511095. doi: 10.1001/jamanetworkopen.2025.11095. PMID 40388166